CLINICAL TRIAL: NCT02243527
Title: Effects of Inspiratory Muscle Training on Respiratory Muscle Mechanics and Haemodynamics in Healthy Adults
Brief Title: Respiratory Muscles and Inspiratory Muscle Training
Acronym: IMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Principal Investigator, Jordan Guenette, Dr. Jordan Guenette, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: H14-00067
Record Dates: First submitted 2014-09-16; First posted 2014-09-18 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-04

CONDITIONS: Respiratory Muscles; Breathing Exercises
Keywords: Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inspiratory Muscle Training (Experimental)
  Interventions: Other: Inspiratory Muscle Training
- Sham-Control Inspiratory Muscle Training (Sham Comparator): Inspiratory muscle training at a low intensity meant to elicit no physiological changes.
  Interventions: Other: Sham Inspiratory Muscle Training

INTERVENTIONS:
Other: Inspiratory Muscle Training — 6-weeks of inspiratory muscle training
  Arms: Inspiratory Muscle Training
Other: Sham Inspiratory Muscle Training — A sham training procedure that is meant to elicit no physiologic changes
  Arms: Sham-Control Inspiratory Muscle Training

SUMMARY:
The effects of inspiratory muscle training (IMT) remain controversial. Many studies have examined the effect IMT has on exercise performance, but any changes to the body that come from IMT have yet to be looked at.

This study will look at how someone breathes can change after IMT. Understanding how IMT changes the body can help us use IMT in different treatments.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally active, 'Moderate' or 'High' category on International Physical Activity Questionnaire Short form questionnaire
* Able to read and understand English
* Pulmonary function within normal limits

Exclusion Criteria:

* History of or currently smoking
* History or current symptoms of cardiopulmonary disease (including asthma and exercise induced asthma)
* Currently participating and training in a sport at a provincial, national, or international level
* Ulcer or tumor in the esophagus, a nasal septum deviation, or recent nasopharyngeal surgery
* Allergies to latex or local anesthetic
* Contraindications to exercise testing

Ages: 19 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2014-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan A Guenette, PhD, Principal Investigator — University of British Columbia/Centre for Heart Lung Innovation
Locations (1):
- Centre for Heart Lung Innovation, Vancouver, British Columbia, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Inspiratory Muscle Training | Sham-Control Inspiratory Muscle Training
Started | 12 | 13
Completed | 12 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inspiratory Muscle Training | Sham-Control Inspiratory Muscle Training | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 13 | 25
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (5) | 24 (4) | 24 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 13 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Diaphragm Electromyography
Description: Using a multipair esophageal electrode catheter we will determine any changes to the electric activity of the diaphragm.
  Diaphragm electromyography (EMG) has been expressed as %max. This unit is determined as the ratio of average EMG value (uV) divided by the maximal EMG activity (uV) generated during a maximal respiratory maneuver (inspiratory capacity during exercise).
Time Frame: Post Intervention - ie. immediately after 5 weeks of inspiratory muscle training
Measure: Mean (Standard Deviation); unit: %max
Arm/Group | Inspiratory Muscle Training | Sham-Control Inspiratory Muscle Training
Number analyzed (Participants) | 12 | 13
%max | 60 (13) | 55 (13)

2. Secondary Outcome: Accessory Respiratory Muscle Activation
Description: Using surface electromyography to determine the activation patterns of accessory respiratory muscles (scalene and sternocleidomastoid).
  Data are expressed as %max. This value is determined by taking the average electromyography (EMG) activity divided by the maximal EMG activity generated during a maximal inspiratory maneuver (inspiratory capacity during exercise).
Time Frame: Post-intervention - ie. immediately after 5 weeks of inspiratory muscle training
Measure: Mean (Standard Deviation); unit: %max
Arm/Group | Inspiratory Muscle Training | Sham-Control Inspiratory Muscle Training
Number analyzed (Participants) | 12 | 13
%max | 10 (7) | 6 (4)

3. Other Pre Specified Outcome: Dyspnoea
Description: Using the modified Borg scale to assess changes in perceived dyspnoea after inspiratory muscle training.
  The modified Borg scale is a 0-10 category ratio scale. The floor (0) of the scale is anchored subjectively to the subjects interpretation of "no breathing discomfort at all", and the ceiling (10) to represent "the most intense breathing discomfort they have experienced or could imagine experiencing".
Time Frame: Post-intervention - ie. immediately after 5 weeks of inspiratory muscle training
Measure: Mean (Standard Deviation); unit: Borg Units
Arm/Group | Inspiratory Muscle Training | Sham-Control Inspiratory Muscle Training
Number analyzed (Participants) | 12 | 13
Borg Units | 8.5 (1.9) | 8.3 (2.5)

4. Other Pre Specified Outcome: Muscle Oxygenation
Description: Using near-infrared spectroscopy to examine if there are any relative changes in concentration (∆umol/Litre) of deoxygenated hemoglobin (HHb) after training. Deoxygenated hemoglobin is used as a surrogate of oxygen extraction specific to the local vasculature of the vastus lateralis,
Time Frame: Post-intervention - ie. immediately after 5 weeks of inspiratory muscle training
Measure: Mean (Standard Deviation); unit: change in umol/Litre HHb
Arm/Group | Inspiratory Muscle Training | Sham-Control Inspiratory Muscle Training
Number analyzed (Participants) | 12 | 13
change in umol/Litre HHb | 15.9 (9.3) | 16.1 (10.3)

ADVERSE EVENTS:
Time Frame: 1 year
Description: No adverse events occurred.
Arm/Group | Inspiratory Muscle Training | Sham-Control Inspiratory Muscle Training
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No